CLINICAL TRIAL: NCT05246020
Title: Efficacy of Neoadjuvant Hyperthermic Intraperitoneal Chemotherapy in Advanced High-grade Serous Ovarian Cancer (the NHIPEC Trial)：a Randomised Controlled Trial
Brief Title: Efficacy of Neoadjuvant Hyperthermic Intraperitoneal Chemotherapy in Advanced High-grade Serous Ovarian Cancer (the NHIPEC Trial)
Acronym: NHIPEC
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2020-KY-050
Record Dates: First submitted 2022-01-24; First posted 2022-02-18 (Actual); Last update posted 2022-02-18 (Actual); Status verified 2022-01

CONDITIONS: Hyperthermic Intraperitoneal Chemotherapy; Neoadjuvant Chemotherapy
Keywords: HIPEC; Neoadjuvant chemotherapy; High-grade serous ovarian cancer
MeSH Terms: interventions — Hyperthermic Intraperitoneal Chemotherapy

STUDY DESIGN:
Intervention Model Description: The eligible patients will be randomised into an experimental group (NHIPEC +intravenous NACT) or a control group (intravenous NACT). Patients in the NHIPEC experimental group will receive NHIPEC and two cycles of intravenous NACT, while patients in the control group will receive three cycles of intravenous NACT. All patients will undergo IDS within 4weeks after the last cycle of NACT.
Who Masked: Outcomes Assessor
Masking Description: All tissue samples harvested during IDS will be subjected to H&E expert pathological evaluation to confirm the diagnosis of high-grade serous ovarian cancer(HGSOC). Omental slides will be independently reviewed by two pathologists to determine those with the greatest amount of viable tumour, and one slide of each site will be selected. The two pathologists, who will be blinded to the written report and each other's results, will independently score each slide according to the CRS system.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NHIPEC (Experimental): Treatment: Four tubes will be placed via the laparoscopic ports and HIPEC will be given within 24 hours after laparoscopic evaluation.
  Interventions: Procedure: HIPEC
- Intravenous NACT (Active Comparator): Drug:Three cycles of intravenous NACT will be given in this group. The regimen of intravenous NACT is docetaxel 60-75mg/m2 followed by carboplatin area under curve(AUC) 5 for a 21-day cycle.
  Interventions: Procedure: intravenous chemotherapy

INTERVENTIONS:
Procedure: HIPEC — Docetaxel (60-75mg/m2) perfusion solution will be infused into the peritoneal cavity through the tubes within 24 hours after the laparoscopic evaluation. Then, perfusate containing cisplatin (75 mg/m2) will be infused 24 hours later. NHIPEC will be administered at 43°C for a duration of 60min. Saline solution (3000mL) will be used to dissolve the drug, and it will be heated and circulated at a flow rate of 300-500 mL/min.
  Arms: NHIPEC
Procedure: intravenous chemotherapy — Patients in the control group will receive three cycles of intravenous NACT. The regimen of intravenous NACT is docetaxel 60-75mg/m2 followed by carboplatin AUC 5 for a 21-day cycle.
  Arms: Intravenous NACT

SUMMARY:
Background: Neoadjuvant chemotherapy (NACT) is an important treatment option for patients with ovarian cancer. Although intravenous NACT can improve optimal resection rates and decrease surgical morbidity and mortality, these advantages do not translate into a survival benefit. Ovarian carcinoma is mainly confined to the peritoneal cavity, which makes it a potential target for hyperthermic intraperitoneal chemotherapy (HIPEC). Our previous study showed that HIPEC could be used in the neoadjuvant setting, which was named neoadjuvant HIPEC (NHIPEC). Since hyperthermia is an excellent chemosensitiser, we hypothesised that the combination of NHIPEC and intravenous NACT could show superior efficacy to intravenous NACT alone. Methods: This study is a single-centre, open-label, randomised (1:1 allocation ratio) phase 2 trial. A total of 80 patients will be randomly assigned into an experimental group (NHIPEC+intravenous NACT) or a control group (intravenous NACT). Patients in the experimental group will receive NHIPEC following laparoscopic evaluation, and four tubes will be placed via the laparoscopic ports, which will be used to administer NHIPEC. Then, perfusion with docetaxel (60-75 mg/m2) will be performed (43°C for 60 min, Day 0) followed by cisplatin (75 mg/m2, Day 1) infusion (43°C for 60 min) 24 hours later. After NHIPEC, two cycles of intravenous NACT will be given. Patients in the control group will receive three cycles of intravenous NACT. The primary endpoint is the proportion of patients who achieve a Chemotherapy Response Score (CRS) of 3 according to the CRS system. The secondary endpoints include progression-free survival, overall survival and the rates of complete resection and NHIPEC-related adverse events.

ELIGIBILITY:
Inclusion Criteria:

1. International Federation of Gynecology and Obstetrics(FIGO) stage IIIC-IVA, HGSOC
2. Patients with Fagotti score ≥8
3. Adequate kidney function (blood creatinine 58-96 µmol/L)
4. Adequate haematological function (haemoglobin ≥110g/L, leucocytes ≥4.0×109/L, neutrophils ≥2.0×109/L, platelets≥100×109/L)
5. Adequate liver function (serum total bilirubin 3.4-22.2µmol/L, alanine aminotransferase (ALT) 7-40U/L, aspartate aminotransferase (AST) 13-35U/L, AST/ALT ≤1.5)
6. World Health Organization(WHO) score 0-2

Exclusion Criteria:

1. Patients who had received chemotherapy, radiotherapy or any kind of targeted therapy.
2. Patients with complete intestine obstruction.
3. Expected life span ≤8 weeks.
4. Complicated with any other known malignancies.
5. Patients with poor cardiopulmonary function, which would limit compliance with study requirements.

Ages: 17 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2020-12-01 (Actual); Primary Completion 2022-12-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
chemotherapy response score(CRS) 3 | At the end of cycle 3 NACT (each cycle is 21 days)
  the proportion of chemotherapy response score 3, which means a better outcome

SECONDARY OUTCOMES:
progression-free survival(PFS) | From date of randomization until the date of first documented progression, assessed up to 3 years
  progression-free survival
overall survival(OS) | From date of randomization until the time of death from any cause, assessed up to 3 years
  overall survival
Rate of R0 resection | At the end of cycle 3 NACT (each cycle is 21 days),when IDS is conducted
  the R0 resection rate of interval debulking surgery(IDS)
NHIPEC-related adverse effects | during the procedure
  the adverse effects of NHIPEC

CONTACTS AND LOCATIONS:
Overall Officials: Jing Li, Doctor, Principal Investigator — Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University
Locations (1):
- Sun Yat-sen Memorial Hospital, Guangzhou, Other (Non U.s.), China

IPD SHARING:
Plan to Share IPD: No
After data publication